CLINICAL TRIAL: NCT02197611
Title: Development of a Specific Measure for Assessing Adherence in Adult Patients With Hemophilia. The Haemo-Adhaesione Questionnaire
Brief Title: Development of a Specific Measure for Assessing Adherence in Adult Patients With Hemophilia.
Acronym: ADHAESIONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, ANA TORRES-ORTUÑO, PhD, Universidad de Murcia
Other Study IDs: Haemo Adhaesione; Haemo-Adhaesione (Other: UMurcia)
Record Dates: First submitted 2014-07-15; First posted 2014-07-22 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Haemophilia
Keywords: Haemophilia; Adherence of Treatment; Knowledge of Illness; Medical-patient Relationship; Illness Behavior; Treatment Difficulties.
MeSH Terms: conditions — Hemophilia A; Illness Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Validation group: Group of patients who we will consult the characteristics of the scale designed and will be made the statistical calculations of validity, reliability and reproducibility

SUMMARY:
Research project for the development, construction and validation of a questionnaire of adherence to treatment in adult patients with hemophilia. It aims to build a scale according to five relevant dimensions of adherence to treatment: 1) physician-patient relationship, 2) knowledge of the disease, 3) previous bleeding problems, 4) knowledge of future consequences and difficulties, and 5) benefits of treatment.

DETAILED DESCRIPTION:
* Descriptive study for the construction of a multidimensional scale of adherence to treatment in adult patients with hemophilia.
* Validation of a scale specific measure for patients with hemophilia that includes 5 dimensions that may affect adherence to treatment: a) the doctor-patient, b) regarding knowledge of the disease, c) the previous hemorrhages, d) knowledge future sequels, e) difficulties with treatment.
* Statistical and psychometric analysis of the adherence questionnaire for adult patients with hemophilia.
* Description of the theoretical framework that justifies the completion of the questionnaire, and the choice of the dimensions and items that make up the measurement scale.
* The questionnaire obtained in this project will identify the actual degree of patient adherence to multidisciplinary treatment, taking as gold standard, compliance with pharmacological treatment (the difference between the treatment prescribed and consumed).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A or B.
* Patients over 18 years of age.

Exclusion Criteria:

* Patients with neurological or cognitive impairments that hinder oral and written comprehension.
* Patients who have not signed the informed consent document

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with haemophilia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Phase substantive for the creation of a scale | Screening visit
  The theoretical framework and objectives for the creation of the scale is created. The questionnaire was developed teóricasdel dimensions and items of each dimension are identified. In this testing phase, the pilot is 5 Hematologists physicians experienced in hemophilia (no contact between them) and a sample of the target population (± 12 patients with hemophilia). The structure of this phase include:
  * Identify and define the theorical framework of customs and attributes.
  * Identification of behaviors that represent the attribute.
  * Test design specifications.
  * Construction of the items.
  * External judgment by judges
  * Discussion with the target population
  * Analysis of item-objective congruence
  * Analysis of the interview with patients and selection of items
  * Selection of an initial set of items
  * Application of the first version and analysis items
  * Selection of items in accordance with standard psychometric
Structural phase for the creation of a scale | Screening visit
  This phase is carried out the questionnaire to a pilot sample (± 50 patients with hemophilia) and the choice of format is made. Similarly, an analysis of differential functioning or bias of the items is performed. The structure of this phase include:
  * Implementation of the final scale
  * Determination of ground and ceiling effect of the scale
  * Analysis of the structure of the scale
  * Identifying relevant dimensions
  * Calculate the reliability
  * Determination of the reproducibility
  * Establishing convergent and discriminant validity
Empirical phase for the creation of a scale | Screening visit
  This phase is carried out applying the scale to a general sample (patient 100-150). After the statistical and convergence and discriminant analysis (other scales) and the study of responsibility (with drug consumption data) will be made. The structure of this phase include:
  * Selecting one or more external criteria
  * To establish concurrent validity
  * Checking empirical hypotheses
  * Determination of responsiveness
  * Study interpretability
  * Design guidelines for the administration and scoring of scales
  * Design cutoff scores

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad de Murcia, Murcia, Murcia, Spain